CLINICAL TRIAL: NCT04684082
Title: Prospective, Single-center, Single-arm, Open-label Observational PMCF Study - Evaluation of Performance and Safety of Colonic Irrigation With the Colon Hydromat as a Non-oral Bowel Preparation for Colonoscopy
Brief Title: Evaluation of Performance and Safety of Colonic Irrigation With the Colon Hydromat as a Non-oral Bowel Preparation for Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herrmann Apparatebau GmbH (Industry)
Collaborators: CERES GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: HRR015CHT
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-12

CONDITIONS: Colonic Irrigation
Keywords: Colon Hydrotherapy; Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Patients will receive colonic irrigation as bowel preparation prior to colonoscopy.
  Interventions: Device: Colonic irrigation with the Colon Hydromat

INTERVENTIONS:
Device: Colonic irrigation with the Colon Hydromat — A designated health professional will administer to the patient the colonic irrigation procedure - using the "Colon Hydromat" device, a CE certified device for colonic irrigation and cleansing before endoscopic procedures.

SUMMARY:
This is a clinical study with a medical device that bears the CE mark (approval for marketing in the EU) and is applied within its intended use. It is a prospective, single-centre, single-arm, open-label, observational post-market clinical follow-up (PMCF) study using the "Colon Hydromat" system for bowel preparation prior to colonoscopy. The patients will be treated according to the clinical routine and in accordance with the current IFU.

Aim of the study is to confirm safety and performance (effectiveness) of colon hydrotherapy as bowel preparation for colonoscopy. Colonic irrigation is regarded as a substitute for standard oral colonic purgative solutions for colonoscopy preparation, especially for patients, who cannot tolerate oral preparations or want to have alternatives because they have experienced the current oral preparations as a burdensome process.

DETAILED DESCRIPTION:
This observational study is intended to answer the question, if the colon hydrotherapy (colonic irrigation with the "Colon Hydromat") works in real-life practice.

Colonic irrigation is regarded as a substitute for standard oral colonic purgative solutions for colonoscopy preparation. The advantage of colonic irrigation is that there is no unpleasant taste, it avoids the discomfort of diarrheic episode and there is no need to drink a large volume of water or fluids. The patient will receive the bowel irrigation with the "Colon Hydromat" directly before colonoscopy, at the same day. Aim of this study is to confirm performance (effectiveness), in terms of an adequate bowel preparation and safety of the "Colon-Hydromat", as alternative bowel cleansing device prior to colonoscopy. The primary performance (effectiveness) endpoint for this study is the colonic cleanliness, defined as overall quality of bowel cleansing as measured by the Boston Bowel Preparation Scale (BBPS). The primary safety endpoints for this study are adverse device events (ADE) and serious adverse device effects (SADE), product and procedure related.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication of colonoscopy: inclusion is considered if patients require a colonoscopy and
* desire an alternative bowel preparation method to standard of oral polyethylene glycol or other orally taken purgatives, or do not tolerate the oral preparations, or had an inadequate colon cleansing following traditional oral preparation, in order to complete the colonoscopy at the same day.
* Adult patients (≥ 18 years old) having signed the informed consent.
* Being able to respond to the self-administered questionnaire.

Exclusion Criteria:

* Psychiatric conditions and inability to provide informed consent
* Emergency colonoscopy
* Off-label use (application is not within the IFU)
* Pregnancy and lactation period
* The patient has one of the contraindications listed in the IFU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (men and women) who are planned for a colonoscopy and where anorectal colonic irrigation with the specula can be performed, will be included into the study.
  The colonic irrigation is regarded as alternative bowel preparation to oral preparations, especially for patients who:
  * cannot tolerate oral preparations (e.g. cannot drink large volumes, nausea, vomiting), or
  * want to have alternatives because they have experienced the current oral preparations as a burdensome process, or
  * had an inadequate colon cleansing following traditional oral preparation, in order to complete the colonoscopy at the same day.
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-02-03 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel preparation (Colonic Cleanliness), evaluated through the Boston Bowel Preparation Scale (BBPS). | day 1
  Quality of bowel preparation validated by numerical scale for bowel cleanse (0-9 best)
Adverse device events (ADE) and collection of SADE (device or procedure related). | day 1
  Assessment of ADE: Patients will be asked in questionnaires, if they had any adverse events, especially nausea, vomiting, pain/cramps, dizziness and headache and rate of patients where colonic irrigation had to be aborted. Assessment of SADE: will be assessed at end of colonoscopy by investigator.

SECONDARY OUTCOMES:
BBPS for each segment. | day 1
  BBPS will be assessed in each bowel segment (left, transverse, right).
Patient satisfaction. | day 1
  Patient satisfaction with respect to convenience and comfort/ discomfort, and preference/acceptance, as evaluated by a questionnaire (questions to the patient; no score).
User satisfaction and usability. | day 1
  User satisfaction and usability, as measured by a questionnaire (questions to the patient; no score).
Details to colonic irrigation. | day 1
  Time taken to complete the colon irrigation with the "Colon Hydromat".
Details to colonic irrigation. | day 1
  Number of cycles used for cleaning the colon.
Details to colonic irrigation. | day 1
  Volume of water used for cleaning the colon.
Colonoscopic findings. | day 1
  Characteristics of all polyps/lesions detected:
  Location (right, transverse, or left colon) and size.
  General assessment of colon anatomy and other circumstances related to the colon:
  No abnormality detected / tortuous / very long/ diverticular disease / stenosis / severe constipation / weak muscle tone of the sphincter - build-up of pressure was insufficient.
Rate of colonoscopy termination. | day 1
  Rate of colonoscopy termination due to inadequate bowel preparation.
Procedure time of colonoscopy. | day 1
  Procedure time of colonoscopy (time from intubation to withdrawal).
Withdrawal time. | day 1
  Withdrawal time: the total time for withdrawal from cecum to anus; this includes all interventions or delays (e.g. biopsies, polypectomies…).
Cecal intubation rate. | day 1
  Cecal intubation rate (reaching the cecum or anastomosis, if present).
Runway time. | day 1
  Time interval between the patient's end of bowel cleaning / colonic irrigation and the moment of colonoscope insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Teich, Prof. Dr. med., Principal Investigator — Study centre Leipzig - Internistic Joint Practice
Locations (1):
- Internistische Gemeinschaftspraxis für Verdauungs- und Stoffwechselerkrankungen, Leipzig, Germany